CLINICAL TRIAL: NCT00649311
Title: Clinical Protocol For A Double-Blind, Randomized, Active- Controlled Comparison Study Of The Antihypertensive Effect Of Eplerenone Versus Losartan In Patients With Mild To Moderate Hypertension
Brief Title: A Study To Evaluate The Efficacy Of Eplerenone Compared With Losartan For The Treatment Of Patients With Mild To Moderate Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment; termination not due to safety reasons.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPLA-0501-072; A6141012
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Eplerenone; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eplerenone group (Experimental)
  Interventions: Drug: eplerenone
- Losartan group (Active Comparator)
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: eplerenone — Eplerenone 50 mg oral film-coated tablet once daily for 8 weeks. If blood pressure was uncontrolled (DBP ≥ 90 mmHg) at Week 4, the dose was increased to eplerenone 100 mg oral film-coated tablet once daily for 4 weeks.
  Arms: Eplerenone group
Drug: Losartan — Losartan 50 mg oral capsule once daily for 8 weeks. If blood pressure was uncontrolled (DBP ≥ 90 mmHg) at Week 4, the dose was increased to losartan 100 mg oral capsule once daily for 4 weeks
  Arms: Losartan group

SUMMARY:
The purpose this study is to compare the efficacy of eplereonone and losartan in patients with mild to moderate hypertension.

DETAILED DESCRIPTION:
This Phase 2 study EPLA-0501-072 (A6141012) was conducted beginning 02 April 2003 and was prematurely terminated due to poor enrollment on 12 September 2003. There were no statistical analyses of efficacy conducted because the numbers of patients enrolled were insufficient for inferential analysis due to the poor enrollment. There were no serious adverse events or deaths reported during the study.

ELIGIBILITY:
Inclusion Criteria:

* History of mild to moderate hypertension, or newly diagnosed hypertension, defined as seDBP ≥90 mmHg and <110 mmHg and seSBP <180 mmHg
* Withdrawal of all previous antihypertensives prior to the single-blind placebo run-in period and the double-blind treatment period

Exclusion Criteria:

* Secondary hypertension (e.g., renal, renovascular, or adrenocortical disease, pheochromocytoma, Cushing's syndrome, primary aldosteronism, iatrogenic), severe hypertension, or malignant hypertension
* The patient cannot withdraw from antihypertensives by any route including diuretics, alpha-blockers, betablockers, calcium channel blockers, ACE-I, ARB, or other medications affecting blood pressure; patients who have stable angina and have not had their nitrate dosage changed within the past three months (i.e., on a stable maintenance dose) are eligible for this study; sildenafil citrate, theophylline, or papaverine must not be taken within 24 hours prior to a clinic visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2003-04; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in seated trough cuff diastolic blood pressure (seDBP) at Week 8 | 8 weeks

SECONDARY OUTCOMES:
Mean change from baseline in seated cuff systolic blood pressure (seSBP) at Week 8 | 8 weeks
Percent of patients meeting the goal BP of DBP <90 mmHg or a reduction of ≥10 mmHg in DBP | 8 weeks
Overall safety and tolerability of all treatments as assessed by change in vital signs, 12-lead electrocardiograms, clinical laboratory tests, and adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Taiwan (2):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EPLA-0501-072&StudyName=A%20Study%20To%20Evaluate%20The%20Efficacy%20Of%20Eplerenone%20Compared%20With%20Losartan%20For%20The%20Treatment%20Of%20Patients%20With%20Mild%20To%20Moderate%20Hyperte